CLINICAL TRIAL: NCT01395238
Title: Enhancing Father's Ability to Support Their Preschool Child
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Grant ended and faculty has left the institution
Sponsor: Queens College, The City University of New York (Other)
Collaborators: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Poline Papoulis, Director ORSP, Queens College, The City University of New York
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1U01CE001653 (NIH)
Record Dates: First submitted 2011-05-23; First posted 2011-07-15 (Estimated); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Fathers; Parenting; High-risk; Child Maltreatment; Prevention
Keywords: fathers; parenting; high-risk; child maltreatment; prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Wait-List Group (No Intervention)
- Parenting Group (Experimental): Experimental Condition. Group-based, 8 weekly sessions/2 hours per week.
  Interventions: Behavioral: Fathers Supporting Success in preschoolers

INTERVENTIONS:
Behavioral: Fathers Supporting Success in preschoolers — Group-based, 8 weekly session for 2.0 hours/week.
  Arms: Parenting Group

SUMMARY:
This study focuses on the development of the Fathers Supporting Success in Preschoolers (FSSP) Program, which combines evidence-based parenting interventions with Dialogic Reading to engage fathers in and improve parenting and child behavior.

ELIGIBILITY:
Inclusion Criteria:

* Male Guardian
* Child enrolled in partnering Head Start site

Exclusion Criteria:

* Mental Health issues that prohibit involvement in group-based prevention study (e.g., psychosis)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2010-09; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Parenting Behavior Checklist | post treatment (8 weeks after start of treatment )
  Reporting change in parenting behavior from baseline to immediately after intervention
Eyberg Child Behavior Inventory | post treatment (8 weeks after start of treatment )
  Reporting change in child behavior from baseline to immediately after intervention

SECONDARY OUTCOMES:
Center for Epidemiological Studies Depression Scale | post treatment (8 weeks after start of treatment )
  Reporting change in paternal depression from baseline to immediately after intervention
Parent Cognition Scale | post treatment (8 weeks after start of treatment )
  Measurement of parents cognitions regarding children behavior. reporting change in parental cognitions from baseline to immediatley after intervention
Preschool Language Scales | post treatment (8 weeks after start of treatment )
  Assessment of child langauge skills. reporting changes in children's language from baseline to immediatley after intervention
Developing Skills Checklist | post treatment (8 weeks after start of treatment )
  Assessment of early literacy skills. Reporting changes in children's literacy skills from baseline to immediately after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Anil Chacko, PhD, Principal Investigator — Queens College, CUNY
Locations (1):
- Queens College, Flushing, New York, United States